CLINICAL TRIAL: NCT05282264
Title: Acceptability of Hybrid Closed-loop Systems in Patients Living With Highly Unbalanced Type 1 Diabetes
Acronym: HCL-VHP
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: IDRCB 2022-A00144-39
Record Dates: First submitted 2022-02-04; First posted 2022-03-16 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-06

CONDITIONS: Type 1 Diabetes
Keywords: Highly unbalanced Type 1 diabetes; hybrid closed loops; acceptability; efficacy and safety; quality of life
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Equipment and Supplies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient with hybrid closed-loop systems
  Interventions: Other: device
- Patient without hybrid closed-loop systems

INTERVENTIONS:
Other: device — closed-loop insulin
  Groups: Patient with hybrid closed-loop systems

SUMMARY:
While closed-loop insulin delivery (CLID) systems demonstrated safety and effectiveness in patients with unbalanced type 1 diabetes (T1D), no studies have included patients with highly and chronically unbalanced diabetes.

The investigators conduct a retrospective, observational, and single-center study to evaluate the acceptability, safety, and efficacy of a CLID system in patients living with T1D (≥2 years) with a HbA1c>11% in the past 12 months and a mean HbA1c >10% over the past three years. Efficacy was assessed using continuous glucose monitoring parameters.

DETAILED DESCRIPTION:
If hybrid closed-loop systems (HCLS) ("artificial pancreas") for automated insulin administration have demonstrated their great interest in patients living with moderately unbalanced type 1 diabetes (T1D) (HbA1c < 8 .6% on average), no study has looked at their safety, acceptability and efficacy in patients living with highly and chronically unbalanced T1D (HbA1c > 11%). These patients, often young, present more or less advanced microangiopathic complications (retinopathy, nephropathy, neuropathy, etc.) or are highly exposed to the appearance of these complications, the prevention of which, whether primary or secondary, involves obtaining a good glycemic balance over time. These patients "escape" the possibilities of current insulin therapy, whether by multiple insulin injections or by insulin pump, more or less coupled to a continuous glucose monitoring system. Automated insulin delivery systems could be a solution to achieve less catastrophic glycemic control in some of these patients. The investigators are proposing a pilot study aimed at evaluating acceptability, safety and effectiveness of a HCLS currently available in France (the SMARTGUARD™ MINIMED™ 780G or the Control-IQ) in patients followed in the diabetology department of the Centre Hospitalier Sud-Francilien (CHSF), living with highly unbalanced T1D (HbA1c > 11%) in the context of usual follow-up.

ELIGIBILITY:
Inclusion Criteria:

Patients with closed loop system :

* Adult patients
* With T1D for at least 2 years
* Follow-up in the diabetes department of the CHSF
* Having a laboratory HbA1c > 11% at least once during the past year and at least one other HbA1c > 10% in the previous 3 years
* Accepting the closed loop system as part of their support
* Subject informed of the study and not objecting to it

Patients without closed loop system :

Adult patients

* With T1D for at least 2 years
* Follow-up in the diabetes department of the CHSF
* Having a laboratory HbA1c > 11% at least once during the past year and at least one other HbA1c > 10% in the previous 3 years
* Refusing the closed loop system as part of their support or
* Patients for whom a multi-professional medical and paramedical collegial discussion (including diabetologist and nurse referents of the patient) within the service leads to the evaluation of an unfavorable benefit/risk ratio
* Subject informed of the study and not objecting to it

Exclusion Criteria:

Patients with closed loop system :

* Patients without an Internet connection, or without a smartphone or computer
* Patients for whom a multi-professional medical and paramedical collegial discussion (including diabetologist and patient referent nurse) within the department results in the assessment of an unfavorable benefit/risk ratio (patients with a history of interrupted pump treatment on medical decision, serious psychiatric disorders…)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed in the diabetes department of the Centre Hospitalier Sud Francilien
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Acceptability of hybrid closed-loop systems | at 12 months
  Maintenance rate of a hybrid closed-loop system in patients living with highly unbalanced T1D (HbA1c > 11%) and followed in the diabetes department of the CHSF

SECONDARY OUTCOMES:
Demographic characteristics : age | at day 0
  year
  * lives alone or not; precariousness index,
  * psychiatric history,
  * number of hospitalizations related to diabetes, severe hypoglycaemia, ketoacidosis in the last 3 years,
  * weight, body mass index (BMI),
  * treatment of diabetes: pump (brand, year), multiple injections (MDI),
  * complications of diabetes; microangiopathic: retinopathy (shape and stage), nephropathy (estimated glomerular filtration rate by the CKD-EPI formula, albuminuria/creatinine ratio), neuropathies; macroangiopathic
  * average HbA1c level for the last 3 years
Demographic characteristics : gender | at day 0
  feminine or masculine
  * psychiatric history,
  * number of hospitalizations related to diabetes, severe hypoglycaemia, ketoacidosis in the last 3 years,
  * weight, body mass index (BMI),
  * treatment of diabetes: pump (brand, year), multiple injections (MDI),
  * complications of diabetes; microangiopathic: retinopathy (shape and stage), nephropathy (estimated glomerular filtration rate by the CKD-EPI formula, albuminuria/creatinine ratio), neuropathies; macroangiopathic
  * average HbA1c level for the last 3 years
Demographic characteristics : level of education | at day 0
  year
Demographic characteristics : currrent activity | at day 0
  student, active, retired, unemployed, etc.
Demographic characteristics : duration of diabete | at day 0
  year
HbA1c | at day 0
  HbA1c
Efficiency | At baseline, 3, 6, and 12 months
  * If the patient has interrupted the treatment with hybrid closed-loop, reason for the discontinuation,
  * % of time spent under HCLS,
  * Change of pump between M0 and M12 (Yes/no).
  * Change of transmitter between M0 and M12 (Yes/no),
  * Average total insulin dose per day,
  * Basal/Bolus ratio,
  * Amount of carbohydrates entered/day,
  * Target objective (mg/dL) set,
  * Number of sensors consumed
  * Number of sensor malfunctions
  * International consensus criteria on the interpretation of continuous glucose monitoring (CGM):
    * Evolution of the time spent in the target (TIR),
    * Change in time above target (TAR) for hyperglycaemia > 250 mg/dL, from 181 to 250 mg/dL,
    * Evolution of the time spent below the target of 54 to 69 mg/dL and < 54 mg/dL,
    * Evolution of the glycemic average,
    * Evolution of the coefficient of variation (CV).
Quality | At baseline, 3, 6, and 12 months
  Questionnaire Diabetes Quality of life : from 1 ( very satisfaying) to 5 (very unsatisfactory)
Patient satisfaction | At baseline, 3, 6, and 12 months
  Questionnaire Diabetes Quality of life : from 3 (many) to -3 (less)
Hypoglycemia Fear | At baseline, 3, 6, and 12 months
  Hypoglycemia Fear Survey : from 0 (never) to 4 (almost always)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Penfornis, Corbeil-Essonnes, Centre Hospitalier Sud Francilien
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Deepchand S, Balla V, Eroukhmanoff J, Ly Sall K, Romain B, Lejeune M, Penfornis A, Amadou C. Closed-Loop Insulin Delivery Systems for People with Type 1 Diabetes and Chronic Very Poor Metabolic Control: It Works and Is Safe! Diabetes Technol Ther. 2024 Feb;26(2):125-129. doi: 10.1089/dia.2023.0379. Epub 2024 Jan 11. PMID 37955849